CLINICAL TRIAL: NCT06769061
Title: The Use of Acupuncture to Reduce Chemotherapy Induced Peripheral Neuropathy (CIPN) in Gynaecological Cancer Patients - a Pilot Randomised Controlled Trial
Brief Title: The Use of Acupuncture to Reduce Chemotherapy Induced Peripheral Neuropathy in Gynaecological Cancer Patients
Acronym: AcuCIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Kar Loen CHAN (Other)
Responsible Party: Sponsor-Investigator, Karen Kar Loen CHAN, Department Chairperson and Clinical Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AcuCIN
Record Dates: First submitted 2024-12-20; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Gynaecological, Urological or Rectal Cancer; Chemotherapy-Induced Peripheral Neuropathy; Acupuncture
Keywords: Gynaecological Cancer; Acupuncture; Chemotherapy induced peripheral neuropathy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Eligible patients will be 1:1:1 randomised to three groups: electroacupuncture group, sham acupuncture group and waiting-list (usual care) control group. For electroacupuncture and sham acupuncture groups, the assessors and the patients will be blinded to the treatment given.
  1. Electroacupuncture group - patients will receive 6 weeks of electroacupuncture, 2 sessions per week, by a qualified TCM practitioner from the School of Chinese Medicine.
  2. Sham acupuncture group - patients will receive 6 weeks of sham acupuncture similar to the above.
  3. Waiting-list (usual care) control group - patients will not receive any treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomised into three groups. Both the subjects (acupuncture and sham acupuncture group) and the gynaecological clinical research team responsible for the clinical care and neuropathy assessments will be blinded. There is no blinding for waiting-list control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupuncture (Experimental): Patients randomised to this arm will receive intervention of electroacupuncture. They will receive 6 weeks of electroacupuncture, 2 sessions per week, 30 min per session.
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator): Patients randomised to this arm will receive sham comparator, sham acupuncture. They will receive 6 weeks of sham acupuncture, 2 sessions per week, 30 min per session.
  Interventions: Device: sham acupuncture
- Waiting-list (usual care) control (No Intervention): Patients randomised to the waiting-list control group will receive standard of care managementf for CIPN.

INTERVENTIONS:
Procedure: Acupuncture — Patients will receive 6 weeks of electroacupuncture, 2 sessions per week, 30 min per session Stainless steel, single-use, sterile, and disposable needles will be used. We will use the bilateral acupoints LI4 (He-Gu), TE5 (Wai-Guan), LI11 (Qu-Chi), and LU5 (Chi-Ze) for upper limbs. For lower limb numbness, we will use the bilateral acupoints of LV3 (Tai-Chong), ST41 (Jie-Xi), SP6 (San-Yin-Jiao), and GB34 (Yang-Ling-Quan) for the numbness of back of feet, or the bilateral acupoints of KI1 (Yong-Quan), KI3 (Tai-Xi), SP6 (San-Yin-Jiao), and GB34 (Yang-Ling-Quan). After skin disinfection, sterile adhesive pads will be placed on bilateral LI4 (Hegu), TE5 (Waiguan), LI11 (Quchi), and LU5 (Chize). Following each needle insertion, acupuncturists will perform equal manipulations of twirling, lifting, and thrusting on the needle by acupuncturists to achieve the de qi sensation. These 4 acupoints (He-Gu, Qu-Chi, San-Yin-Jiao, Yang-Ling-Quan) will be electrically stimulated for 30 min.
  Arms: Acupuncture
Device: sham acupuncture — Patients will receive 6 weeks of sham acupuncture, 2 sessions per week, 30 min per session. The Streitberger sham acupuncture needle designed specifically for sham acupuncture trials will be used. Patients will feel the needle on the skin, but the needle actually will not puncture the skin. These 4 acupoints (He-Gu, Qu-Chi, San-Yin-Jiao, Yang-Ling-Quan) will be connected to the electrical stimulation device KWD-808I MULTI-PURPOSE Health device (Great Wall Company), but not stimulated. The needle will remain for 30 minutes. without stimulating the acupoints. The sham acupuncture will be used within the trocar. The trocar will be fixed by a base on the skin with sticker. The trocar-base-sticker will be used for both acupuncture group and sham acupuncture control group, so they are exactly the same in appearance. Patients cannot see if there is acupuncture or sham acupuncture within the trocar.
  Arms: Sham acupuncture

SUMMARY:
Objectives:

To explore the feasibility and effectiveness of acupuncture on reducing Chemotherapy Induced Peripheral Neuropathy (CIPN) in gynaecological cancer patients who have received carboplatin and paclitaxel chemotherapy combination. Results of this pilot trial will provide preliminary information for a potential a larger scale multicentre study.

Hypothesis:

Acupuncture can significantly reduce CIPN in gynaecological cancer patients treated with chemotherapy

Design and subjects:

This is a pilot, prospective randomised controlled trial. This is an exploratory trial to evaluate the feasibility and effectiveness of acupuncture in reducing CIPN in gynaecological cancer patients. Eligible patients will be 1:1:1 randomised to three groups: electroacupuncture group, sham acupuncture group and waiting-list (usual care) control group. For electroacupuncture and sham acupuncture groups, the assessors and the patients will be blinded to the treatment given.

1. Electroacupuncture group - patients will receive 6 weeks of electroacupuncture, 2 sessions per week, by a qualified Traditional Chinese Medicine practitioner from the School of Chinese Medicine.
2. Sham acupuncture group - patients will receive 6 weeks of sham acupuncture similar to the above.
3. Waiting-list (usual care) control group - patients will not receive any treatment.

Main outcomes:

Acupuncture effects will be assessed at baseline and 3, 6,12 weeks post intervention by:

1. Patient reported outcome measures: FACT/GOG-Ntx questionnaire for assessing CIPN symptoms and EORTC-QLQ-C30 and CIPN20 questionnaires for assessing quality of life symptom
2. Clinician reported outcome measures: NCI-CTCAE grading for CIPN by clinicians and Semmes-Weinstein monofilament test as an objective measurement of CIPN.

Data analysis:

Intention to treat analysis will be carried out. Baseline demographics will be compared between the 3 groups. Change from baseline total score will be calculated and analysed using 2-sample t-test. 95% CI will be reported for treatment differences. Score for different subcategories will be analysed in a similar manner. Data collected at week 6 will be used for outcome analysis. P<0.05 will be considered as statistically significant. Acupuncture efficacy, effectiveness and placebo effect will be indicated by comparison of acupuncture vs. sham acupuncture, acupuncture vs. waiting-list, and sham acupuncture vs. waiting-list, respectively.

Expected results: Patients in the acupuncture arm will have reduced numbness and peripheral neuropathy and improved quality of life without any adverse event.

DETAILED DESCRIPTION:
Subjects will be recruited by research assistant at the gynaecological oncology clinics at Queen Mary Hospital. All potential subjects will be required to fill in a screening questionnaire to assess the degree of neuropathy. Screening blood test (Complete blood picture) will be taken within 1 month of starting acupuncture. Eligible subjects will be enrolled into the study according to the inclusion and exclusion criteria. Any type of acupuncture or message in daily Traditional Chinese Medicine clinic will be prohibited during the trial once the subject is enrolled.

Subjects will be allocated to the 3 groups through computer generated randomization: acupuncture, sham acupuncture or the waiting-list (usual care) control group on a 1:1:1 ratio. Allocations will be kept within sealed opaque envelopes. Once a patient has been enrolled, an envelope is opened and the patient is then offered the allocated treatment regimen. Both the subjects (acupuncture and sham acupuncture group) and the gynaecological clinical research team responsible for the clinical care and neuropathy assessments will be blinded to the results.

Patients who are randomised to sham acupuncture or waiting-list control group will be offered the option of receiving 12 acupuncture treatments when they finish all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Diagnosis of uterine (endometrial) cancer, ovarian cancer and cervical cancer
* ECOG=0-2
* Life expectancy of > 6 months
* Completed at least 6 cycles of carboplatin or cisplatin chemotherapy together with paclitaxel at least 3 months before joining the study
* Able to read and understand the questionnaires
* PNQ score of C or above

Exclusion Criteria:

* Bleeding tendency
* Abnormal clotting profile
* Platelet lower than 50
* Received acupuncture in the past
* Currently receiving chemotherapy treatment
* Known neurological disorders or pre-existing neuropathy unrelated to chemotherapy
* Routinely take aspirin or any anticoagulant drugs
* Having active skin infection
* With pacemaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 75 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy Induced Peripheral Neuropathy associated quality of life measured by Functional Assessment of Cancer Therapy / Gynecologic Oncology Group - Neurotoxicity subscale (FACT/GOG-NTX) total score | From enrollment to 6 weeks after end of treatment including: baseline at enrollment, after 3 weeks of treatment/enrollment, after 6 weeks of treatment (end of treatment)/ enrollment, and 6 weeks after end of treatment /12 weeks after enrollment
  This questionnaire provides a targeted assessment of peripheral neuropathy symptoms. It consists of a total of 38 items on physical, social, emotional and functioning well-being with 11 questions focusing on neurotoxicity. This instrument is validated and has been used in Phase 3 clinical trials. The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
The changes in quality of life assessed by European Organisation For Research And Treatment Of Cancer-Quality of Life-C30 (EORTC-QLQ-C30) questionnaires | From enrollment to 6 weeks after end of treatment including: baseline at enrollment, after 3 weeks of treatment/enrollment, after 6 weeks of treatment (end of treatment)/ enrollment, and 6 weeks after end of treatment /12 weeks after enrollment
  Quality of life will be assessed by patient reported EORTC-QLQ-C30 questionnaires): C30 is a well validated instrument to assess quality of life in cancer patients. It consists of 30 items encompassing physical, emotional, social and functional aspects. Higher scores indicate better quality of life
The changes in quality of life assessed by European Organisation For Research And Treatment Of Cancer-Quality of Life-Chemotherapy Induced Peripheral Neuropathy 20 (EORTC-QLQ-CIPN20) questionnaires | From enrollment to 6 weeks after end of treatment including: baseline at enrollment, after 3 weeks of treatment/enrollment, after 6 weeks of treatment (end of treatment)/ enrollment, and 6 weeks after end of treatment /12 weeks after enrollment
  Quality of life will be assessed by patient reported EORTC-QLQ-CIPN20 questionnaires: CIPN20 is a 20 items additional module to EORTC-QLQ-C30 focusing on Chemotherapy Induced Peripheral Neuropathy symptoms. Higher scores indicate better quality of life
assess the changes in light touch sensation by Semmes-Weinstein filaments test | From enrollment to 6 weeks after end of treatment including: baseline at enrollment, after 3 weeks of treatment/enrollment, after 6 weeks of treatment (end of treatment)/ enrollment, and 6 weeks after end of treatment /12 weeks after enrollment
  For assessment the light touch sensation, the research assistant will perform Semmes-Weinstein filaments (SWM) test at the same time points as the patient's questionnaires (Baseline, Week 3, 6, 12). Each monofilament will be used for three consecutive times on the same point, and the participants are asked to provide information about their sense of touch with their eyes closed. The testing session starts using the thinnest monofilament, moving to a thicker one if the participant does not feel a monofilament.
assess the safety by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) grading | From enrollment to 6 weeks after end of treatment including: baseline at enrollment, after 3 weeks of treatment/enrollment, after 6 weeks of treatment (end of treatment)/ enrollment, and 6 weeks after end of treatment /12 weeks after enrollment
  Any adverse effects and their severity during treatment procedures including dizziness, nausea, vomiting, pain, discomfort, sweating, palpitations, bleeding and bruising will be assessed by CTCAE. The intervention will be discontinued if patients suffer from any serious adverse events (AEs). AE will be managed according to standard of care procedures.
assess the chemotherapy induced peripheral pain in numeric rating scale | From enrollment to 6 weeks after end of treatment including: baseline at enrollment, after 3 weeks of treatment/enrollment, after 6 weeks of treatment (end of treatment)/ enrollment, and 6 weeks after end of treatment /12 weeks after enrollment
  Numeric rating scale represents a key element for measuring pain intensity and symptomatology. It ranges from 0 to 10. 0 means no pain and 10 means maximum pain.
Explore the acupuncture expectancy by Acupuncture expectancy scale (for acupuncture and sham acupuncture group) | At baseline and week 3 (after receiving treatment for 3 weeks)
  In order to control the bias from placebo effect of acupuncture, acupuncture expectance scale will be used to measure the patients' expectations of positive outcomes from the treatment. It is a validated measurement with four items, with score ranging from 4 to 20
Explore the acupuncture credibility by Acupuncture credibility questionnaire (for acupuncture and sham acupuncture group) | At week 3 (after receiving treatment for 3 weeks)
  Acupuncture credibility questionnaire is a questionnaire to control the bias from different patients' credibility of acupuncture practitioners. It is a validated assessment including 4 questions with score ranging from 0 to 6. 0 means minimum and 6 means maximum agreement of the item
Changes in inflammatory biomarkers | From enrollment to end of treatment including: baseline at enrollment, after 6 weeks of treatment (end of treatment)/ enrollment
  Changes in inflammatory biomarkers after acupuncture will be explored. The BD cytometric Bead Array system (CBA) will be used to quantify the level of inflammation panel (IL10, IL12-p70, IL1β, IL6), Th1/Th2 panel (IL2, IL4, IL5, TNF, IFNγ), B cell activation panel (CD79b, BLNK, Btk, Syk, PLCγ), T cell activation panel (TCRz, SLP-76, ZAP70, Pyk2, Itk), and the Complements panel (C4a, C3a, C5a). The plasma level of CRP will be determined by ELISA assay. Fecal samples will be sent for fecal sequencing and profiling to explore the potential mechanisms of acupuncture effects.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kar Loen Prof CHAN, MBBChir (Cantab); MD (HK), Principal Investigator — Department of Obstetrics and Gynaecology, the University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No